CLINICAL TRIAL: NCT05767762
Title: Evertor Muscle Activity as a Predictor of Achilles Tenotomy Before 1 Year in the Management of Idiopathic Varus Equinus Clubfoot
Brief Title: Evertor Muscle Activity as a Predictor of Achilles Tenotomy in the Management of Idiopathic Varus Equinus Clubfoot
Acronym: PBVE-Muscle
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Lenval (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 22-HPNCL-09
Record Dates: First submitted 2023-03-02; First posted 2023-03-14 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-03

CONDITIONS: Clubfoot
Keywords: Muscle activity; scale; Achilles tenotomy
MeSH Terms: conditions — Clubfoot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Idiopathic Clubfoot (Experimental)
  Interventions: Other: scale Idiopathic Clubfoot

INTERVENTIONS:
Other: scale Idiopathic Clubfoot — The Dimeglo and the muscle activity scale will be performed at 3, 6 and 12 months with patient with idiopathic clubfoot

SUMMARY:
Clubfoot is an orthopedic congenital malformation of the lower limb of the newborn evaluated by the Dimeglio score. There is a deficit of muscular balance between the agonists and antagonists to the deformity. The Dimeglio score takes into account the muscular activity but only up to one point out of 20. This study proposes to use a muscle scale inspired by the Dimeglio score to see if there is a correlation between muscle activity and the risk of tenotomy before 1 year. It will also assess the inter-examiner reproducibility of this scale.

This study is a prospective cohort study with a duration of 8 years to include about 100 feet. Infants with idiopathic Clubfoot treated with the functional method at up to 15 days of life will be included. Feet will be assessed at an inclusion visit and then at 3-6-12 months.

The primary endpoint will be the need for Achilles tenotomy before 1 year of age. The secondary endpoint will be inter-examiner reproducibility determined by statistical analysis.

The expectation of this study would be to define a predictive factor of the evolution of the PBVE in order to refine the treatment earlier.

DETAILED DESCRIPTION:
Clubfoot is a congenital orthopedic deformity of the lower limb in newborns. It is characterized by a triple deformity of the foot: equinus, supination and adduction of the forefoot. It can be bilateral or unilateral. PBVE can be idiopathic or associated with another etiology such as neurological, rheumatological, etc.

There is a muscular hypoplasia of the muscles antagonistic to the PBVE and an imbalance of force between the agonists and antagonists to the benefit of the deformity. There is also an abnormality of the fibular and posterior tibial nerves.

The aim of the study is the muscular evaluation of the PBVE. The scientific literature is relatively poor on the subject. In the first year of life, if the articular evaluation of the PBVE is very precise, the muscular scoring seems less well taken into account. In the Dimeglio score, the muscular criterion counts for 1 point (against 16 articular points) if it is possible to obtain a muscular contraction of the antagonists. It does not specify which muscles are present nor the active reducibility of the deformity. A scale based on the Dimeglio score has been created to evaluate muscle activity. To fill it out, the practitioner will have to stimulate the muscles antagonistic to the deformity by tactile stimulation.

This will be an 8-year prospective cohort study that will look for a correlation between the muscle deficit and the risk of tenotomy before 1 year as well as the quality of inter-examiner reproduction of the scale. This duration is necessary to obtain a sufficient number of inclusions (100 feet).

Infants with idiopathic Clubfoot treated with the functional method at up to 15 days of life will be included. At the first consultation, we will perform the Dimeglio score and our muscle activity scale. The Dimeglio and the muscle activity scale will be performed at 3, 6 and 12 months. The population included will need to be sufficient to ensure that all levels of muscle scoring are represented.

The primary endpoint will be the need for Achilles tenotomy before 1 year. The secondary endpoint will be inter-examiner reproducibility determined by statistical analysis.

The expectation of this study would be to define a predictive factor of the evolution of the PBVE in order to refine the treatment earlier.

ELIGIBILITY:
Inclusion Criteria:

* idiopathic clubfoot, managed by the functional method, managed before D15 to perform the initial assessment.

Exclusion Criteria:

* syndromic clubfoot, management other than functional method, management after D15

Ages: 0 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2023-04-26 (Actual); Primary Completion 2031-03 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Surgery | maximum 1 year after inclusion
  number of patient who need for Achilles tenotomy

SECONDARY OUTCOMES:
Inter-examiner reproducibility | through study completion, an average of 8 years
  measure with statistical study the Inter-examiner reproducibility

CONTACTS AND LOCATIONS:
Locations (1):
- Hopitaux Pediatriques de Nice Chu-Lenval, Nice, France